CLINICAL TRIAL: NCT02161406
Title: A Phase 2 Study to Evaluate Subcutaneous Abatacept vs. Placebo in Diffuse Cutaneous Systemic Sclerosis- a Double-blind, Placebo-controlled, Randomized Controlled Trial.
Brief Title: A Study of Subcutaneous Abatacept to Treat Diffuse Cutaneous Systemic Sclerosis
Acronym: ASSET
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dinesh Khanna, MD, MS (Other)
Collaborators: Bristol-Myers Squibb (Industry); National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor-Investigator, Dinesh Khanna, MD, MS, Associate Professor of Rheumatology/ Internal Medicine, University of Michigan
Organization: University of Michigan (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IM101-344; 1UM1AI110557 (NIH)
Record Dates: First submitted 2014-06-03; First posted 2014-06-11 (Estimated); Results first posted 2019-06-18 (Actual); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Diffuse Cutaneous Systemic Sclerosis
Keywords: Scleroderma
MeSH Terms: conditions — Scleroderma, Diffuse | interventions — Abatacept

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Abatacept (Active Comparator): 125 mg SC abatacept vs SC placebo administered weekly for 12 months, with a 24-week open-label extension
  Interventions: Drug: Abatacept
- Placebo (Placebo Comparator): 125mg Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Abatacept — Subjects will be treated with injections of 125 mg of abatacept or placebo weekly for 52 weeks
  Other Names: Orencia
  Arms: Abatacept
Drug: Placebo — 125 mg of Placebo
  Arms: Placebo

SUMMARY:
The study hypothesis is that SC abatacept is safe and shows evidence of efficacy (improvement in modified Rodnan score [mRSS]) in patients with diffuse cutaneous systemic sclerosis (dcScc) compared to matching placebo.

DETAILED DESCRIPTION:
This study is a randomized placebo-controlled double-blind phase 2 trial of patients with dcSSc. Eligible participants will be randomized in a 1:1 ratio to either 125 mg SC abatacept or matching placebo, stratified by duration of dcSSc disease duration (<18 months vs >18 to </=36 months). Study participants will be treated for 12 months on double-blind study medication, followed by an additional 24 weeks of open-label SC abatacept therapy. 86 patients will be randomized in approximately 35 centers in the US, Canada and Europe, with the goal of analyzing 74 participants. The investigators study will test whether abatacept is statistically superior to placebo in reducing the MRSS at month 12 and explore the ability of abatacept to prevent or reverse progression in patients with early disease duration and lower MRSS scores, and reverse established disease in patients with longer disease duration and higher MRSS scores.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of Systematic Sclerosis (SSc), as defined using the 2013 American College of Rheumatology/ European Union League Against Rheumatism classification of SSc
2. Diffuse Systemic Sclerosis (dcSSc) as defined by LeRoy and Medsger
3. Disease duration of ≤ 36 months (defined as time from the first non-Raynaud phenomenon manifestation)
4. For disease duration of ≤ 18 months: ≥ 10 and ≤ 35 mRSS units at the screening visit
5. For disease duration of >18-36 months: ≥ 15 and ≤ 45 mRSS units at the screening visit and one of the following:

   * Increase ≥ 3 in mRSS units compared with the last visit within previous 1-6 months
   * Involvement of one new body area with ≥ 2 mRSS units compared with the last visit within the previous 1-6 months
   * Involvement of two new body areas with ≥ 1 mRSS units compared with the last visit within the previous 1-6 months
   * Presence of 1 or more Tendon Friction Rub
6. Age ≥ 18 years at the screening visit
7. If female of childbearing potential, the patient must have a negative pregnancy test at screening and baseline visits
8. Oral corticosteroids (≤ 10 mg/day of prednisone or equivalent) and NSAIDs are permitted if the patient is on a stable dose regimen for

   * 2 weeks prior to and including the baseline visit.
9. ACE inhibitors, calcium-channel blockers, proton-pump inhibitors, and/or oral vasodilators are permitted if the patient is on a stable dose for ≥ 2 weeks prior to and including the baseline visit.

Exclusion Criteria:

1. Rheumatic disease other than dcSSc; it is acceptable to include patients with fibromyalgia and scleroderma-associated myopathy
2. Limited cutaneous systemic sclerosis or sine scleroderma at the screening visit
3. Major surgery (including joint surgery) within 8 weeks prior to screening visit
4. Infected ulcer prior to randomization
5. Treatment with any investigational agent within ≤ 4 weeks (or 5 half-lives of the investigational drug, whichever is longer) of the baseline visit
6. Previous treatment with cell-depleting therapies, including investigational agents, including but not limited to, CAMPATH, anti-CD4, anti-CD5, anti-CD3, anti-CD19, and ABA
7. Anti-CD20, and cyclophosphamide within 12 months prior to baseline visit.
8. Use of Intravenous Immunoglobulin (IVIG) within 12 weeks prior to baseline visit
9. Previous treatment with chlorambucil, bone marrow transplantation, or total lymphoid irradiation
10. Immunization with a live/attenuated vaccine within ≤ 4 weeks prior to the baseline visit
11. Treatment with methotrexate, hydroxychloroquine, cyclosporine A, azathioprine, mycophenolate mofetil rapamycin, colchicine, or D-penicillamine, within≤ 4 weeks prior to the baseline visit
12. Treatment with etanercept within ≤ 2 weeks, infliximab, certolizumab, golimumab, ABA or adalimumab within ≤ 8 weeks, anakinra within ≤ 1 week prior to the baseline visit
13. Pulmonary disease with FVC ≤ 50% of predicted, or DLCO (uncorrected for hemoglobin ) ≤ 40% of predicted at the screening visit
14. Pulmonary arterial hypertension (PAH) as determined by right heart catheterization or on PAH approved medications for PAH. It is acceptable to use PDFE-5 inhibitors for Raynaud's and digital ulcers.
15. Subjects at risk for tuberculosis (TB). Specifically excluded from this study will be participants with a history of active TB within the last 3 years, even if it was treated; a history of active TB greater than 3 years ago, unless there is documentation that the prior anti-TB treatment was appropriate in duration and type; current clinical, radiographic, or laboratory evidence of active TB; and latent TB that was not successfully treated (≥ 4 weeks).
16. Positive for hepatitis B surface antigen prior to the baseline visit
17. Positive for hepatitis C antigen, if the presence of hepatitis C virus was also shown with polymerase chain reaction or recombinant immunoblot assay prior to baseline visit
18. Subjects at risk for tuberculosis (TB). Specifically excluded from this study will be participants with a history of active TB within the last 3 years, even if it was treated; a history of active TB greater than 3 years ago, unless there is documentation that the prior anti-TB treatment was appropriate in duration and type; current clinical, radiographic, or laboratory evidence of active TB; and latent TB that was not successfully treated (≥ 4 weeks).
19. Any of the following at the screening visit: Hemoglobin <8.5 g/dL; WBC < 3,000/mm3 (<3 x 109/L); platelets < 100,000/mm3 (<3 x 109/L); serum creatinine > 2 x ULN; serum ALT or AST > 2 x ULN
20. Severe skin thickening (mRSS 3) on the inner aspects of thighs, upper arms, or abdomen
21. Patients with a history of anaphylaxis to abatacept

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2018-09-12 (Actual); Study Completion 2018-10-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dinesh Khanna, MD, MS, Principal Investigator — University of Michigan
Locations (27):
- United States (23):
  - Arthritis Associates of Southern California, Los Angeles, California
  - University of California- Los Angeles, Los Angeles, California
  - Stanford University, Redwood City, California
  - Georgetown University, Washington D.C., District of Columbia
  - Northwestern University, Chicago, Illinois
  - Harvard Mass General, Boston, Massachusetts
  - Boston University, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Rutgers University Clinical Research Center, New Brunswick, New Jersey
  - Steffens Scleroderma Center, Albany, New York
  - NorthWell Health, Great Neck, New York
  - Hospital for Special Surgery, New York, New York
  - Columbia University, New York, New York
  - Cleveland Clinic, Cleveland, Ohio
  - Ohio State University Medical Center, Columbus, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - University of Texas Health Center at Houston, Houston, Texas
  - University of Utah, Salt Lake City, Utah
  - Swedish Health Services, Seattle, Washington
- Canada (3):
  - St. Joseph Health Care London, London, Ontario
  - Mount Sinai Hospital, Toronto, Ontario
  - Jewish General Hospital, Montreal, Quebec
- Royal Free Hospital, London, United Kingdom

REFERENCES:
- [Derived] Mehta BK, Espinoza ME, Franks JM, Yuan Y, Wang Y, Wood T, Gudjonsson JE, Spino C, Fox DA, Khanna D, Whitfield ML. Machine-learning classification identifies patients with early systemic sclerosis as abatacept responders via CD28 pathway modulation. JCI Insight. 2022 Dec 22;7(24):e155282. doi: 10.1172/jci.insight.155282. PMID 36355434
- [Derived] Chung L, Spino C, McLain R, Johnson SR, Denton CP, Molitor JA, Steen VD, Lafyatis R, Simms RW, Kafaja S, Frech TM, Hsu V, Domsic RT, Pope JE, Gordon JK, Mayes MD, Sandorfi N, Hant FN, Bernstein EJ, Chatterjee S, Castelino FV, Ajam A, Allanore Y, Matucci-Cerinic M, Whitfield ML, Distler O, Singer O, Young A, Nagaraja V, Fox DA, Furst DE, Khanna D. Safety and efficacy of abatacept in early diffuse cutaneous systemic sclerosis (ASSET): open-label extension of a phase 2, double-blind randomised trial. Lancet Rheumatol. 2020 Dec;2(12):e743-e753. doi: 10.1016/S2665-9913(20)30237-X. Epub 2020 Oct 19. PMID 34966900
- [Derived] Khanna D, Spino C, Johnson S, Chung L, Whitfield ML, Denton CP, Berrocal V, Franks J, Mehta B, Molitor J, Steen VD, Lafyatis R, Simms RW, Gill A, Kafaja S, Frech TM, Hsu V, Domsic RT, Pope JE, Gordon JK, Mayes MD, Schiopu E, Young A, Sandorfi N, Park J, Hant FN, Bernstein EJ, Chatterjee S, Castelino FV, Ajam A, Wang Y, Wood T, Allanore Y, Matucci-Cerinic M, Distler O, Singer O, Bush E, Fox DA, Furst DE. Abatacept in Early Diffuse Cutaneous Systemic Sclerosis: Results of a Phase II Investigator-Initiated, Multicenter, Double-Blind, Randomized, Placebo-Controlled Trial. Arthritis Rheumatol. 2020 Jan;72(1):125-136. doi: 10.1002/art.41055. Epub 2019 Dec 10. PMID 31342624
- See also: To learn more about the Scleroderma program at the University of Michigan — http://www.med.umich.edu/scleroderma

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Abatacept | Placebo
Started | 44 | 44
Completed | 34 | 35
Not Completed | 10 | 9
Not completed — Death | 2 | 1
Not completed — Lost to Follow-up | 2 | 1
Not completed — Withdrawal by Subject | 2 | 4
Not completed — investigator withdrew subject | 3 | 1
Not completed — Lack of Efficacy | 1 | 1
Not completed — relocation | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety population includes all of the randomized participants who received at least one dose of study medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | Abatacept | Placebo | Total
Number analyzed (Participants) | 44 | 44 | 88
Age, Continuous [Mean (Standard Deviation); unit: years] | 50 (12) | 49 (13) | 49 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 35 | 66
  Male | 13 | 9 | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 7 | 11
  Not Hispanic or Latino | 40 | 36 | 76
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 3 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 3 | 6
  White | 35 | 37 | 72
  More than one race | 4 | 0 | 4
  Unknown or Not Reported | 0 | 1 | 1
Disease Duration [Mean (Standard Deviation); unit: years] — Disease duration for this outcome is defined as the disease duration since the first non-Raynaud's sign or symptom until the screening visit.
  years | 1.66 (0.84) | 1.52 (0.79) | 1.59 (0.81)
dcSSc Disease Duration <= 18 months [Count of Participants; unit: Participants] — dcSSc disease duration is defined as the time from the diagnosis of diffuse cutaneous systemic sclerosis (dcSSc) until screening.
  Participants | 26 | 27 | 53
mRSS [Mean (Standard Deviation); unit: units on a scale] — modified Rodnan skin scores (mRSS) have a range from 0 to 51, with higher score indicating greater severity of systemic scleroderma
  units on a scale | 23.34 (7.947) | 21.57 (7.328) | 22.45 (7.652)
FVC% Predicted [Mean (Standard Deviation); unit: percent predicted] — FVC is Forced vital capacity, a measure of lung function. FVC % Predicted is calculated using equations from Hankinson [Hankinson JL, Odencrantz JR, Fedan KB. Spirometric reference values from a sample of the general U.S. population. Am J Respir Crit Care Med. 1999;159(1):179-87], incorporating age, gender, and race. It is calculated as the (FVC Observed / FVC predicted) * 100, where FVC predicted is calculated relative to a reference population.
  percent predicted | 84.19 (13.504) | 86.49 (16.597) | 85.34 (15.087)
DLCO% Predicted, Corrected for Hemoglobin [Mean (Standard Deviation); unit: percent predicted] — Percent predicted diffusing capacity for carbon monoxide (DLCO), corrected for hemoglobin (Hb), is reported. For adult males, the equation (expressing Hb in gm•dL-1) is DLCO predicted × (1.7*Hb / (10.22+Hb)). In adult women, the equation is DLCO predicted × (1.7*Hb / (9.38+Hb)). Percent predicted DLCO was entered directly into the eCRFs, based on equipment and testing techniques meeting ATS/ERS requirements (Crapo RO, Morris AH. Standardized single breath normal values for carbon monoxide diffusing capacity. Am.Rev.Respir.Dis 1981;123:185-189).
  percent predicted | 79.57 (18.117) | 76.45 (18.439) | 78.01 (18.241)
Patient Global Assessment [Mean (Standard Deviation); unit: units on a scale] — Patient global assessment for overall disease represents the patient's assessment of the patient's global scleroderma on a 0 (excellent) -10 (extremely poor) Likert scale.
  units on a scale | 3.88 (2.206) | 4.31 (2.561) | 4.09 (2.384)
HAQ-DI [Mean (Standard Deviation); unit: units on a scale] — HAQ-DI is the Health Assessment Question Disability Index that assesses the extent of a patient's functional ability. The HAQ-DI overall score ranges from 0 (no disability) to 3 (severe disability).
  units on a scale | 1.14 (0.716) | 0.97 (0.701) | 1.05 (0.710)
Physician Global Assessment [Mean (Standard Deviation); unit: units on a scale] — Physician global assessment for overall disease: This assessment represents the physician's assessment of the patient's current disease activity on a 0 (excellent) -10 (extremely poor) Likert scale.
  units on a scale | 4.77 (1.669) | 4.76 (1.665) | 4.77 (1.657)
Proportion of Participants with >= 1 Tendon Friction Rubs [Count of Participants; unit: Participants] — Tendon friction rubs in systemic sclerosis have been associated with diffuse cutaneous skin disease, increased disability and poor survival. They were considered present if palpable on physical exam in the shoulder, elbow, wrist, metacarpophalangeal (MCP) joint, knee, and ankle. We report the proportion of subjects with at least one tendon friction rub.
  Participants | 19 | 13 | 32
Proportion of Participants with >= 1 Large Joint Contractures [Count of Participants; unit: Participants] — Joint contractures are recognized by the loss of joint motion upon physical exam. We report the proportion of subjects with at least one large joint contracture.
  Participants | 31 | 32 | 63
Swollen Joint Count [Mean (Standard Deviation); unit: number of swollen joints] — 28 joints are assessed for swelling (positive or negative). The number of swollen joint count ranges from 0 to 28.
  number of swollen joints | 3.64 (5.620) | 3.86 (5.849) | 3.75 (5.704)
Proportion of Participants with >= 1 Swollen Joint Count [Count of Participants; unit: Participants] — 28 joints are assessed for swelling (positive or negative). The number of swollen joint count ranges from 0 to 28. We report the proportion of participants with >= 1 swollen joint.
  Participants | 21 | 21 | 42
Proportion of Participants with Previous Use of Immunosuppressives [Count of Participants; unit: Participants] | 12 | 5 | 17
Proportion of Participants with Previous Use of Prednisone [Count of Participants; unit: Participants] | 12 | 5 | 17

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants With at Least One Adverse Events (AEs) or Serious AEs (SAEs) in 1 Year
Description: Safety is measured using AEs, including clinical significant changes in vital signs, laboratory test abnormalities and clinical tolerability of abatacept, and using serious AEs
Time Frame: 52 weeks
Population: mITT population includes all of the randomized participants who received at least one dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Abatacept | Placebo
Number analyzed (Participants) | 44 | 44
Participants | 35 | 40

2. Primary Outcome: Change From Baseline in the Modified Rodnan Skin Score (mRSS) to Month 12
Description: The efficacy of treatment on skin fibrosis will be measured by changes from baseline to month 12 in mRSS, a measure of skin thickness. mRSS scores have a range from 0 to 51, with higher score indicating greater severity of SSc (worse outcome).
Time Frame: Baseline and 52 weeks
Population: mITT population includes all of the randomized participants who received at least one dose of study medication.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Abatacept | Placebo
Number analyzed (Participants) | 44 | 44
units on a scale | -6.24 (1.14) | -4.49 (1.14)
Statistical Analysis 1: Comparison: Abatacept vs Placebo; Test type: Superiority; p = 0.28, Mixed Models Analysis

3. Secondary Outcome: Change From Baseline to Month 12 in Patient Global Assessment for Overall Disease
Description: Patient global assessment for overall disease represents the patient's assessment of the patient's global scleroderma on a 0 (excellent) -10 (extremely poor) Likert scale. Higher score means worse outcome.
Time Frame: Baseline and Week 52
Population: mITT population includes all of the randomized participants who received at least one dose of study medication.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Abatacept | Placebo
Number analyzed (Participants) | 44 | 44
score on a scale | -0.31 (0.423) | -0.09 (0.457)
Statistical Analysis 1: Comparison: Abatacept vs Placebo; Test type: Superiority; p = 0.73, Mixed Models Analysis

4. Secondary Outcome: Change From Baseline to Month 12 in Physician Global Assessment for Overall Disease
Description: This assessment represents the physician's assessment of the patient's current disease activity on a 0 (excellent) -10 (extremely poor) Likert scale. Higher score means worse outcome.
Time Frame: Baseline and Week 52
Population: mITT population includes all of the randomized participants who received at least one dose of study medication.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Abatacept | Placebo
Number analyzed (Participants) | 44 | 44
score on a scale | -1.3 (0.290) | -0.35 (0.318)
Statistical Analysis 1: Comparison: Abatacept vs Placebo; Test type: Superiority; p = 0.03, Mixed Models Analysis

5. Secondary Outcome: Change in % Predicted FVC
Description: FVC is Forced vital capacity, a measure of lung function. FVC % Predicted is calculated using equations from Hankinson [Hankinson JL, Odencrantz JR, Fedan KB. Spirometric reference values from a sample of the general U.S. population. Am J Respir Crit Care Med. 1999;159(1):179-87], incorporating age, gender, and race. It is calculated as the (FVC Observed / FVC predicted) * 100, where FVC predicted is calculated relative to a reference population.
Time Frame: Baseline and 52 weeks
Population: mITT population includes all of the randomized participants who received at least one dose of study medication.
Measure: Least Squares Mean (Standard Error); unit: percent predicted
Arm/Group | Abatacept | Placebo
Number analyzed (Participants) | 44 | 44
percent predicted | -1.34 (1.24) | -4.13 (1.22)
Statistical Analysis 1: Comparison: Abatacept vs Placebo; Test type: Superiority; p = 0.11, Mixed Models Analysis

6. Secondary Outcome: Change From Baseline to Month 12 in FVC (in ml)
Description: FVC = forced vital capacity, a measure of lung function
Time Frame: Baseline and Week 52
Population: mITT population includes all of the randomized participants who received at least one dose of study medication.
Measure: Least Squares Mean (Standard Error); unit: ml
Arm/Group | Abatacept | Placebo
Number analyzed (Participants) | 44 | 44
ml | -36.39 (43.82) | -121.6 (46.39)
Statistical Analysis 1: Comparison: Abatacept vs Placebo; Test type: Superiority; p = 0.19, Mixed Models Analysis

7. Secondary Outcome: Change From Baseline to Month 12 in HAQ-DI - Overall
Description: The HAQ-DI is the Health Assessment Question Disability Index that assesses the extent of a patient's functional ability. The HAQ-DI overall score ranges from 0 (no disability) to 3 (severe disability). Higher score means worse outcome.
Time Frame: Baseline and Week 52
Population: mITT population includes all of the randomized participants who received at least one dose of study medication.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Abatacept | Placebo
Number analyzed (Participants) | 44 | 44
score on a scale | -0.17 (0.07) | 0.11 (0.07)
Statistical Analysis 1: Comparison: Abatacept vs Placebo; Test type: Superiority; p = 0.005, Mixed Models Analysis

8. Secondary Outcome: Change From Baseline to Month 12 in SHAQ-DI VAS - Overall Disease
Description: Scleroderma-Health Assessment Question Disability Index visual analogue scales (VAS) assess the burden of digital ulcers, Raynaud's, gastrointestinal involvement, breathing, and overall disease. The VAS scale for disease severity ranges from 0 (no disease) to 150 (very severe). A higher score means a worse outcome.
Time Frame: Baseline and Week 52
Population: mITT population includes all of the randomized participants who received at least one dose of study medication.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Abatacept | Placebo
Number analyzed (Participants) | 44 | 44
score on a scale | -7.42 (5.638) | 3.52 (6.045)
Statistical Analysis 1: Comparison: Abatacept vs Placebo; Test type: Superiority; p = 0.19, Mixed Models Analysis

9. Secondary Outcome: Change From Baseline to Month 12 in SHAQ-DI VAS - Breathing
Description: Scleroderma-Health Assessment Question Disability Index visual analogue scales (VAS) assess the burden of digital ulcers, Raynaud's, gastrointestinal involvement, breathing, and overall disease. The VAS scale for how much breathing problems interfered with daily activities ranges from 0 (do not limit activities) to 150 (very severe limitation). A higher score means a worse outcome.
Time Frame: Baseline and Week 52
Population: mITT population includes all of the randomized participants who received at least one dose of study medication.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Abatacept | Placebo
Number analyzed (Participants) | 44 | 44
score on a scale | 9.30 (5.51) | 16.95 (5.85)
Statistical Analysis 1: Comparison: Abatacept vs Placebo; Test type: Superiority; p = 0.34, Mixed Models Analysis

10. Secondary Outcome: Change From Baseline to Month 12 in SHAQ-DI VAS - Raynaud's
Description: Scleroderma-Health Assessment Question Disability Index visual analogue scales (VAS) assess the burden of digital ulcers, Raynaud's, gastrointestinal involvement, breathing, and overall disease. The VAS scale for how much Raynaud's interfered with daily activities ranges from 0 (does not limit activities) to 150 (very severe limitation). A higher score means a worse outcome.
Time Frame: Baseline and Week 52
Population: mITT population includes all of the randomized participants who received at least one dose of study medication.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Abatacept | Placebo
Number analyzed (Participants) | 44 | 44
score on a scale | 7.58 (6.60) | -3.64 (7.17)
Statistical Analysis 1: Comparison: Abatacept vs Placebo; Test type: Superiority; p = 0.25, Mixed Models Analysis

11. Secondary Outcome: Change From Baseline to Month 12 in SHAQ-DI VAS - Burden of Digital Ulcers
Description: Scleroderma-Health Assessment Question Disability Index visual analogue scales (VAS) assess the burden of digital ulcers, Raynaud's, gastrointestinal involvement, breathing, and overall disease. The VAS scale for how much finger ulcers interfered with daily activities ranges from 0 (do not limit activities) to 150 (very severe limitation). A higher score means a worse outcome.
Time Frame: Baseline and Week 52
Population: mITT population includes all of the randomized participants who received at least one dose of study medication.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Abatacept | Placebo
Number analyzed (Participants) | 44 | 44
score on a scale | -3.18 (5.13) | 8.67 (5.52)
Statistical Analysis 1: Comparison: Abatacept vs Placebo; Test type: Superiority; p = 0.12, Mixed Models Analysis

12. Secondary Outcome: Change From Baseline to Month 12 in SHAQ-DI VAS - GI Involvement
Description: Scleroderma-Health Assessment Question Disability Index visual analogue scales (VAS) assess the burden of digital ulcers, Raynaud's, gastrointestinal involvement, breathing, and overall disease. The VAS scale for how much intestinal problems interfered with daily activities ranges from 0 (do not limit activities) to 150 (very severe limitation). A higher score means a worse outcome.
Time Frame: Baseline and Week 52
Population: mITT population includes all of the randomized participants who received at least one dose of study medication.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Abatacept | Placebo
Number analyzed (Participants) | 44 | 44
score on a scale | 9.98 (6.00) | 8.01 (6.42)
Statistical Analysis 1: Comparison: Abatacept vs Placebo; Test type: Superiority; p = 0.82, Mixed Models Analysis

13. Secondary Outcome: Change From Baseline to Month 12 in Swollen Joint Count
Description: 28 joints are assessed for swelling (positive or negative). The number of swollen joint count ranges from 0 to 28. A higher number indicates worse outcome.
Time Frame: Baseline and 52 weeks
Population: mITT population includes all of the randomized participants who received at least one dose of study medication.
Measure: Least Squares Mean (Standard Error); unit: number of swollen joints
Arm/Group | Abatacept | Placebo
Number analyzed (Participants) | 44 | 44
number of swollen joints | -0.11 (0.595) | -0.86 (0.601)
Statistical Analysis 1: Comparison: Abatacept vs Placebo; Test type: Superiority; p = 0.37, Mixed Models Analysis

14. Secondary Outcome: Change From Baseline to Month 12 in Tender Joint Counts
Description: 28 joints are assessed for tenderness (positive or negative). The number of tender joint counts ranges from 0 to 28. A higher number indicates worse outcome.
Time Frame: Baseline and 52 weeks
Population: mITT population includes all of the randomized participants who received at least one dose of study medication.
Measure: Least Squares Mean (Standard Error); unit: number of tender joints
Arm/Group | Abatacept | Placebo
Number analyzed (Participants) | 44 | 44
number of tender joints | -0.71 (0.90) | -1.47 (0.91)
Statistical Analysis 1: Comparison: Abatacept vs Placebo; Test type: Superiority; p = 0.55, Mixed Models Analysis

15. Secondary Outcome: Change From Baseline to Month 12 in PROMIS-29 - Physical Function
Description: The Patient-Reported Outcomes Measurement Information System (PROMIS) 29-item short-form health-reported quality of life measures (PROMIS-29) were administered. The transformed score (T-score) for the physical function domain was used, where 50 (10) is the mean (standard deviation) of a relevant reference population. Higher scores equals more of the concept being measured (i.e., better outcome).
Time Frame: Baseline and Week 52
Population: mITT population includes all of the randomized participants who received at least one dose of study medication.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Abatacept | Placebo
Number analyzed (Participants) | 44 | 44
score on a scale | -1.54 (0.65) | -0.17 (0.69)
Statistical Analysis 1: Comparison: Abatacept vs Placebo; Test type: Superiority; p = 0.15, Mixed Models Analysis

16. Secondary Outcome: Change From Baseline to Month 12 in PROMIS-29 - Anxiety
Description: The Patient-Reported Outcomes Measurement Information System (PROMIS) 29-item short-form health-reported quality of life measures (PROMIS-29) were administered. The transformed score (T-score) for the anxiety domain was used, where 50 (10) is the mean (standard deviation) of a relevant reference population. Higher scores equals more of the concept being measured (i.e., worse outcome).
Time Frame: Baseline and Week 52
Population: mITT population includes all of the randomized participants who received at least one dose of study medication.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Abatacept | Placebo
Number analyzed (Participants) | 44 | 44
score on a scale | -3.5 (1.31) | -1.09 (1.37)
Statistical Analysis 1: Comparison: Abatacept vs Placebo; Test type: Superiority; p = 0.21, Mixed Models Analysis

17. Secondary Outcome: Change From Baseline to Month 12 in PROMIS-29 - Depression
Description: The Patient-Reported Outcomes Measurement Information System (PROMIS) 29-item short-form health-reported quality of life measures (PROMIS-29) were administered. The transformed score (T-score) for the depression domain was used, where 50 (10) is the mean (standard deviation) of a relevant reference population. Higher scores equals more of the concept being measured (i.e., worse outcome).
Time Frame: Baseline and Week 52
Population: mITT population includes all of the randomized participants who received at least one dose of study medication.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Abatacept | Placebo
Number analyzed (Participants) | 44 | 44
score on a scale | -0.02 (1.13) | -0.41 (1.20)
Statistical Analysis 1: Comparison: Abatacept vs Placebo; Test type: Superiority; p = 0.81, Mixed Models Analysis

18. Secondary Outcome: Change From Baseline to Month 12 in PROMIS 29 - Fatigue
Description: The Patient-Reported Outcomes Measurement Information System (PROMIS) 29-item short-form health-reported quality of life measures (PROMIS-29) were administered. The transformed score (T-score) for the fatigue domain was used, where 50 (10) is the mean (standard deviation) of a relevant reference population. Higher scores equals more of the concept being measured (i.e., worse outcome).
Time Frame: Baseline and Week 52
Population: mITT population includes all of the randomized participants who received at least one dose of study medication.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Abatacept | Placebo
Number analyzed (Participants) | 44 | 44
score on a scale | -0.65 (1.29) | -0.98 (1.36)
Statistical Analysis 1: Comparison: Abatacept vs Placebo; Test type: Superiority; p = 0.86, Mixed Models Analysis

19. Secondary Outcome: Change From Baseline to Month 12 in PROMIS-29 - Sleep Disturbance
Description: The Patient-Reported Outcomes Measurement Information System (PROMIS) 29-item short-form health-reported quality of life measures (PROMIS-29) were administered. The transformed score (T-score) for the sleep disturbance domain was used, where 50 (10) is the mean (standard deviation) of a relevant reference population. Higher scores equals more of the concept being measured (i.e.,worse outcome).
Time Frame: Baseline and Week 52
Population: mITT population includes all of the randomized participants who received at least one dose of study medication.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Abatacept | Placebo
Number analyzed (Participants) | 44 | 44
score on a scale | -0.31 (0.57) | -0.21 (0.62)
Statistical Analysis 1: Comparison: Abatacept vs Placebo; Test type: Superiority; p = 0.91, Mixed Models Analysis

20. Secondary Outcome: Change From Baseline to Month 12 in PROMIS-29 - Pain Interference
Description: The Patient-Reported Outcomes Measurement Information System (PROMIS) 29-item short-form health-reported quality of life measures (PROMIS-29) were administered. The transformed score (T-score) for the pain interference domain was used, where 50 (10) is the mean (standard deviation) of a relevant reference population. Higher scores equals more of the concept being measured (i.e., worse outcome).
Time Frame: Baseline and Week 52
Population: mITT population includes all of the randomized participants who received at least one dose of study medication.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Abatacept | Placebo
Number analyzed (Participants) | 44 | 44
score on a scale | -4.10 (1.13) | -1.56 (1.22)
Statistical Analysis 1: Comparison: Abatacept vs Placebo; Test type: Superiority; p = 0.13, Mixed Models Analysis

21. Secondary Outcome: Change From Baseline to Month 12 in PROMIS-29 - Ability to Participate in Social Roles & Activities
Description: The Patient-Reported Outcomes Measurement Information System (PROMIS) 29-item short-form health-reported quality of life measures (PROMIS-29) were administered. The transformed score (T-score) for the ability to participate in social roles and activities domain was used, where 50 (10) is the mean (standard deviation) of a relevant reference population. Higher scores equals more of the concept being measured (i.e., better outcome).
Time Frame: Baseline and Week 52
Population: mITT population includes all of the randomized participants who received at least one dose of study medication.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Abatacept | Placebo
Number analyzed (Participants) | 44 | 44
score on a scale | -1.11 (1.07) | -1.26 (1.14)
Statistical Analysis 1: Comparison: Abatacept vs Placebo; Test type: Superiority; p = 0.92, Mixed Models Analysis

22. Secondary Outcome: Change From Baseline to Month 12 in PROMIS-29 - Pain Intensity
Description: The Patient-Reported Outcomes Measurement Information System (PROMIS) 29-item short-form health-reported quality of life measures (PROMIS-29) were administered. The transformed score (T-score) for the pain intensity domain was used, where 50 (10) is the mean (standard deviation) of a relevant reference population. Higher scores equals more of the concept being measured (i.e., worse outcome).
Time Frame: Baseline and Week 52
Population: mITT population includes all of the randomized participants who received at least one dose of study medication.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Abatacept | Placebo
Number analyzed (Participants) | 44 | 44
score on a scale | -0.72 (0.32) | -0.18 (0.33)
Statistical Analysis 1: Comparison: Abatacept vs Placebo; Test type: Superiority; p = 0.24, Mixed Models Analysis

23. Secondary Outcome: Change From Baseline to Month 12 in SCTC GIT - Composite Score
Description: The SCTC GIT is the UCLA Scleroderma Clinical Trial Consortium Gastrointestinal Instrument. It assesses scleroderma-related gastrointestinal symptoms. The composite score ranges from 0 to 2.83; 0 indicates better health and higher score indicates worse health.
Time Frame: Baseline and Week 52
Population: mITT population includes all of the randomized participants who received at least one dose of study medication.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Abatacept | Placebo
Number analyzed (Participants) | 44 | 44
score on a scale | 0.07 (0.047) | -0.05 (0.050)
Statistical Analysis 1: Comparison: Abatacept vs Placebo; Test type: Superiority; p = 0.07, Mixed Models Analysis

24. Secondary Outcome: ACR CRISS at 12 Months
Description: The American College of Rheumatology Combined Response Index in Systemic Sclerosis is a composite endpoint. It is determined in a 2-step process. The first step assesses whether the patient has had a significant decline in renal or cardiopulmonary involvement. If none of these apply, the second step assesses the probability of improvement by measuring changes in five outcomes and integrating them into a single number using an equation described in Khanna D, Berrocal VJ, et al. [The American College of Rheumatology Provisional Composite Response Index for Clinical Trials in Early Diffuse Cutaneous Systemic Sclerosis. Arthritis and Rheumatology. 2016; 68(2):299-311.]. It incorporates changes in the modified Rodnan skin score, percent predicted forced vital capacity (FVC), patient and physician global assessments, and SHAQ-DI over 1 year. The score ranges from 0 to 1; a higher score indicates better outcome.
Time Frame: Week 52
Population: mITT population includes all of the randomized participants who received at least one dose of study medication.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Abatacept | Placebo
Number analyzed (Participants) | 44 | 44
units on a scale | 0.72 [.005 to .994] | 0.02 [0 to 0.750]
Statistical Analysis 1: Comparison: Abatacept vs Placebo; Test type: Superiority; p = 0.03, van Elteren test; The van Elteren test adjusted for duration of dcSSc. Multiple imputation was used to address missing follow-up data in 5 components of CRISS

25. Secondary Outcome: Change From Baseline to Month 12 in PROMIS - Fatigue
Description: The Patient-Reported Outcomes Measurement Information System (PROMIS) 8-question short-form health-reported quality of life measure fatigue domain was administered. The transformed score (T-score) was used, where 50 (10) is the mean (standard deviation) of a relevant reference population. Higher scores equals more of the concept being measured (i.e., worse outcome).
Time Frame: Baseline and Week 52
Population: mITT population includes all of the randomized participants who received at least one dose of study medication.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Abatacept | Placebo
Number analyzed (Participants) | 44 | 44
score on a scale | -2.44 (1.209) | -0.05 (1.285)
Statistical Analysis 1: Comparison: Abatacept vs Placebo; Test type: Superiority; p = 0.1769, Mixed Models Analysis

26. Secondary Outcome: Change From Baseline to Month 12 in PROMIS - Sleep Disturbance
Description: The Patient-Reported Outcomes Measurement Information System (PROMIS) 4-question short-form health-reported quality of life measure sleep disturbance domain was administered. The transformed score (T-score) was used, where 50 (10) is the mean (standard deviation) of a relevant reference population. Higher scores equals more of the concept being measured (i.e., better outcome).
Time Frame: Baseline and Week 52
Population: Modified Intent-to-Treat population includes all of the randomized participants who received at least one dose of study medication
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Abatacept | Placebo
Number analyzed (Participants) | 44 | 44
score on a scale | -0.31 (0.573) | -0.21 (0.620)
Statistical Analysis 1: Comparison: Abatacept vs Placebo; Test type: Superiority; p = 0.9075, Mixed Models Analysis

27. Secondary Outcome: Change From Baseline to Month 12 in PROMIS - Sleep Impairment
Description: The Patient-Reported Outcomes Measurement Information System (PROMIS) 8-question short-form health-reported quality of life measure sleep impairment domain was administered. The transformed score (T-score) was used, where 50 (10) is the mean (standard deviation) of a relevant reference population. Higher scores equals more of the concept being measured (i.e., worse outcome).
Time Frame: Baseline and Week 52
Population: as for outcome 26
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Abatacept | Placebo
Number analyzed (Participants) | 44 | 44
score on a scale | 0.46 (1.267) | -0.54 (1.320)
Statistical Analysis 1: Comparison: Abatacept vs Placebo; Test type: Superiority; p = 0.5831, Mixed Models Analysis

28. Secondary Outcome: Change From Baseline to Month 12 in HAQ-DI - Dressing and Grooming
Description: The HAQ-DI is the Health Assessment Question Disability Index that assesses the extent of a patient's functional ability. The HAQ-DI subscore ranges from 0 (no disability) to 3 (severe disability). A higher score means worse outcome.
Time Frame: Baseline and Week 52
Population: mITT population includes all of the randomized participants who received at least one dose of study medication.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Abatacept | Placebo
Number analyzed (Participants) | 44 | 44
score on a scale | -0.25 (0.115) | 0.14 (0.119)
Statistical Analysis 1: Comparison: Abatacept vs Placebo; Test type: Superiority; p = 0.0193, Mixed Models Analysis

29. Secondary Outcome: Change From Baseline to Month 12 in HAQ-DI - Hygiene
Description: as for outcome 28
Time Frame: Baseline and Week 52
Population: mITT population includes all of the randomized participants who received at least one dose of study medication.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Abatacept | Placebo
Number analyzed (Participants) | 44 | 44
score on a scale | -0.08 (0.125) | 0.40 (0.132)
Statistical Analysis 1: Comparison: Abatacept vs Placebo; Test type: Superiority; p = 0.0097, Mixed Models Analysis

30. Secondary Outcome: Change From Baseline to Month 12 in HAQ-DI - Arising
Description: as for outcome 28
Time Frame: Baseline and Week 52
Population: mITT population includes all of the randomized participants who received at least one dose of study medication.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Abatacept | Placebo
Number analyzed (Participants) | 44 | 44
score on a scale | -0.23 (0.103) | 0.04 (0.109)
Statistical Analysis 1: Comparison: Abatacept vs Placebo; Test type: Superiority; p = 0.0751, Mixed Models Analysis

31. Secondary Outcome: Change From Baseline to Month 12 in HAQ-DI - Reach
Description: as for outcome 28
Time Frame: Baseline and Week 52
Population: mITT population includes all of the randomized participants who received at least one dose of study medication.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Abatacept | Placebo
Number analyzed (Participants) | 44 | 44
score on a scale | -0.12 (0.176) | 0.03 (0.127)
Statistical Analysis 1: Comparison: Abatacept vs Placebo; Test type: Superiority; p = 0.4927, Mixed Models Analysis

32. Secondary Outcome: Change From Baseline to Month 12 in HAQ-DI - Eating
Description: as for outcome 28
Time Frame: Baseline and Week 52
Population: mITT population includes all of the randomized participants who received at least one dose of study medication.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Abatacept | Placebo
Number analyzed (Participants) | 44 | 44
score on a scale | -0.22 (0.118) | 0.02 (0.122)
Statistical Analysis 1: Comparison: Abatacept vs Placebo; Test type: Superiority; p = 0.1604, Mixed Models Analysis

33. Secondary Outcome: Change From Baseline to Month 12 in HAQ-DI - Grip
Description: as for outcome 28
Time Frame: Baseline and Week 52
Population: mITT population includes all of the randomized participants who received at least one dose of study medication.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Abatacept | Placebo
Number analyzed (Participants) | 44 | 44
score on a scale | -0.29 (0.142) | -0.22 (0.149)
Statistical Analysis 1: Comparison: Abatacept vs Placebo; Test type: Superiority; p = 0.7281, Mixed Models Analysis

34. Secondary Outcome: Change From Baseline to Month 12 in HAQ-DI - Walking
Description: as for outcome 28
Time Frame: Baseline and Week 52
Population: mITT population includes all of the randomized participants who received at least one dose of study medication.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Abatacept | Placebo
Number analyzed (Participants) | 44 | 44
score on a scale | -0.02 (0.100) | 0.18 (0.106)
Statistical Analysis 1: Comparison: Abatacept vs Placebo; Test type: Superiority; p = 0.1679, Mixed Models Analysis

35. Secondary Outcome: Change From Baseline to Month 12 in HAQ-DI - Common Daily Activities
Description: as for outcome 28
Time Frame: Baseline and Week 52
Population: mITT population includes all of the randomized participants who received at least one dose of study medication.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Abatacept | Placebo
Number analyzed (Participants) | 44 | 44
score on a scale | -0.09 (0.113) | 0.08 (0.121)
Statistical Analysis 1: Comparison: Abatacept vs Placebo; Test type: Superiority; p = 0.2906, Mixed Models Analysis

ADVERSE EVENTS:
Time Frame: 52 weeks
Description: Coding of adverse events into body system was performed by the study chair for adverse events and by the medical monitors for serious adverse events.
Arm/Group | Abatacept | Placebo
All-Cause Mortality (participants affected / at risk) | 2/44 | 1/44
Serious Adverse Events (participants affected / at risk) | 9/44 | 12/44
Other Adverse Events (participants affected / at risk) | 35/44 | 40/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Abatacept (N=44) | Placebo (N=44)
Cellulitis of right elbow (Infections and infestations) | 1 (1) | 0 (0)
Healthcare associated pneumonia (HCAP) (Infections and infestations) | 0 (0) | 1 (1)
Left side mastoiditis/ abrythnitis (Infections and infestations) | 1 (1) | 0 (0)
Paronychia (Infections and infestations) | 0 (0) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Atrial Flutter (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1)
Congestive Heart Failure (Cardiac disorders) | 0 (0) | 1 (1)
Digital Ischemia (Cardiac disorders) | 0 (0) | 1 (1)
NSTEMI Myocardial Infarction (Cardiac disorders) | 0 (0) | 1 (1)
Pulmonary Arterial Hypertension (Cardiac disorders) | 0 (0) | 1 (1)
Pulmonary Arterial Hypertension and Pericardial Effusion (Cardiac disorders) | 0 (0) | 1 (1)
Worsening AV block (Cardiac disorders) | 0 (0) | 1 (1)
Anemia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Cholecystitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dysphagia due to GI dysmotility (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dysphagia from myositis and prolonged hospitalization (Gastrointestinal disorders) | 1 (1) | 0 (0)
Erosive esophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
GAVE; Severe anemia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Melena (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pseudo obstruction of the small bowel, paralytic ileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
GAVE (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Depression with Suicidal Ideation (Psychiatric disorders) | 0 (0) | 1 (1)
Basal cell carcinoma (BCC) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Squamous Cell Carcinoma In-situ Left Anterior Ear (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Renal crisis (Renal and urinary disorders) | 3 (3) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Abatacept (N=44) | Placebo (N=44)
Other Non-serious Adverse Events (General disorders) | 13 (23) | 12 (16) — Specific adverse event terms that occurred in < 5% of subjects were pooled.
Other Non-serious Adverse Events (Blood and lymphatic system disorders) | 0 (0) | 3 (3) — Specific adverse event terms that occurred in < 5% of subjects were pooled.
Other Non-serious Adverse Events (Infections and infestations) | 17 (24) | 22 (39) — Specific adverse event terms that occurred in < 5% of subjects were pooled.
Other Non-serious Adverse Events (Musculoskeletal and connective tissue disorders) | 18 (25) | 17 (23) — Specific adverse event terms that occurred in < 5% of subjects were pooled.
Other Non-serious Adverse Events (Nervous system disorders) | 7 (7) | 7 (9) — Specific adverse event terms that occurred in < 5% of subjects were pooled.
Other Non-serious Adverse Events (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 13 (15) — Specific adverse event terms that occurred in < 5% of subjects were pooled.
Other Non-serious Adverse Events (Skin and subcutaneous tissue disorders) | 7 (8) | 7 (12) — Specific adverse event terms that occurred in < 5% of subjects were pooled.
Other Non-serious Adverse Events (Renal and urinary disorders) | 1 (1) | 5 (6) — Specific adverse event terms that occurred in < 5% of subjects were pooled.
Other Non-serious Adverse Events (Cardiac disorders) | 3 (4) | 5 (5) — Specific adverse event terms that occurred in < 5% of subjects were pooled.
Other Non-serious Adverse Events (Endocrine disorders) | 3 (3) | 1 (1) — Specific adverse event terms that occurred in < 5% of subjects were pooled.
Other Non-serious Adverse Events (Ear and labyrinth disorders) | 2 (2) | 1 (1) — Specific adverse event terms that occurred in < 5% of subjects were pooled.
Other Non-serious Adverse Events (Gastrointestinal disorders) | 11 (17) | 13 (18) — Specific adverse event terms that occurred in < 5% of subjects were pooled.
Other Non-serious Adverse Events (Hepatobiliary disorders) | 1 (1) | 4 (4) — Specific adverse event terms that occurred in < 5% of subjects were pooled.
Anemia (Blood and lymphatic system disorders) | 4 (4) | 2 (3)
Diarrhea (Gastrointestinal disorders) | 4 (4) | 6 (6)
Dysphagia (Gastrointestinal disorders) | 3 (3) | 2 (2)
Nausea (Gastrointestinal disorders) | 4 (4) | 4 (5)
Vomiting (Emesis) (Gastrointestinal disorders) | 3 (3) | 2 (2)
Fatigue (General disorders) | 2 (2) | 6 (7)
Weight Loss (General disorders) | 3 (3) | 2 (2)
Upper Respiratory Infection (Infections and infestations) | 3 (3) | 9 (11)
Urinary Tract Infection (Infections and infestations) | 2 (2) | 4 (4)
Headache (Nervous system disorders) | 1 (1) | 6 (8)
Pruritis (Itching) (Skin and subcutaneous tissue disorders) | 4 (4) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2015-12-08): https://cdn.clinicaltrials.gov/large-docs/06/NCT02161406/Prot_000.pdf
  • Statistical Analysis Plan (2018-04-06): https://cdn.clinicaltrials.gov/large-docs/06/NCT02161406/SAP_001.pdf